CLINICAL TRIAL: NCT05507489
Title: A Randomized Controlled Multicenter Clinical Study on the Effectiveness of Jinzhen Oral Liquid in Treating Children With Novel Coronavirus Infection
Brief Title: Clinical Trial of Jinzhen Oral Liquid in Treating Children With COVID-19 Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JZ-2022-nCoV-0.1
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: COVID-19; Child, Only
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): Jinzhen oral liquid(for 3 years old, 10 ml once, twice a day; for 4 to 7 years old, 10 ml a time, 3 times a day; for 8 to 18 years old, 15 ml a time, 3 times a day)
  Interventions: Drug: Jinzhen oral liquid or Jinhuaqinggan granules
- control group (Active Comparator): The usage and dosage of Jinhua Qinggan granules were determined by the researcher according to the patient's condition and recorded truthfully
  Interventions: Drug: Jinzhen oral liquid or Jinhuaqinggan granules

INTERVENTIONS:
Drug: Jinzhen oral liquid or Jinhuaqinggan granules — Jinzhen oral liquid, for 3 years old, 10 ml once, twice a day; for 4 to 7 years old, 10 ml a time, 3 times a day; for 8 to 18 years old, 15 ml a time, 3 times a day.The dosage and usage of Jinhua Qinggan granules were determined by the researcher according to the patient's condition. The drugs were medicated for 14 days.

SUMMARY:
Jinzhen oral liquid and Jinhuaqinggan Granules were used in the treatment and the control group for 14 days, respectively, to evaluate the effect of Jinzhen oral liquid in treating children with novel coronavirus infection.

DETAILED DESCRIPTION:
To evaluate the effect of Jinzhen oral liquid in treating children with novel coronavirus infection by shortening the time of first negative turn of virus, improving clinical symptoms and shortening hospital stay, and to observe the safety of Jinzhen oral liquid in clinical application.A total of 240 Patients aged 3 to 18 years old or asymptomatic infected persons who meet the diagnostic criteria for novel coronavirus infection in the COVID-19 Diagnosis and Treatment Protocol (Trial Version 9)were planned to be enrolled. Jinzhen oral liquid was used in the treatment group, and Jinhuaqinggan Granules was used in the control group, with 120 patients in each group. The subjects took the medication for 14 days (the medication could be stopped in advance if they reached the discharge criteria), and were followed up for 14 days after discontinuation. During the treatment period, the subjects' vital signs, chest imaging examination, novel coronavirus nucleic acid test, blood routine, urine routine, liver and kidney function, and condition and symptoms should be monitored on the follow-up day specified in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* 1. Meet the diagnostic criteria of novel coronavirus infected patients in COVID-19 Diagnosis and Treatment Protocol (Trial Version 9);

  2. Asymptomatic infection or clinical classification of mild or common type;

  3. Aged from 3 to 18 years;

  4. The informed consent process was in accordance with the regulations, and the legal guardian or the children (≥8 years old) signed the informed consent form.

Exclusion Criteria:

* 1. Meet the severe/critical early warning indicators;

  2. Children who used proprietary Chinese medicine of the same type for more than 3 days before enrollment;

  3. Children with diarrhea.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-03-18 (Actual); Primary Completion 2022-09-10 (Estimated); Study Completion 2023-03-17 (Estimated)

PRIMARY OUTCOMES:
First negative time of COVID-19 | up to 6 months
  First negative time of COVID-19

SECONDARY OUTCOMES:
Clinical symptom disappearance rate/time | up to 6 months
  Clinical symptom disappearance rate/time
The hospitalization time | up to 6 months
  The hospitalization time
Incidence of conversion to severe/critical illness Incidence of conversion to severe/critical illness Incidence of conversion to severe/critical illness | up to 6 months
  Incidence of conversion to severe/critical illness

CONTACTS AND LOCATIONS:
Locations (1):
- Phase I Clinical Research Center, Qingdao, Shandong, China